CLINICAL TRIAL: NCT00000912
Title: A Phase II, Randomized Trial of Amprenavir as Part of Dual Protease Inhibitor Regimens (Placebo-Controlled) in Combination With Abacavir, Efavirenz, and Adefovir Dipivoxil Versus Amprenavir Alone in HIV-Infected Subjects With Prior Exposure to Approved Protease Inhibitors and Loss of Virologic Suppression as Reflected by a Plasma HIV-1 RNA Concentration >= 1,000 Copies/ml
Brief Title: A Study on Amprenavir in Combination With Other Anti-HIV Drugs in HIV-Positive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 398; 11354 (Registry Identifier: DAIDS ES); Substudy ACTG 5003s
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Placebos; Drug Therapy, Combination; HIV Protease Inhibitors; VX 478; Anti-HIV Agents; Viral Load; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; abacavir; amprenavir; Nelfinavir; efavirenz; Carnitine; adefovir dipivoxil; Saquinavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Levocarnitine
Drug: Adefovir dipivoxil
Drug: Saquinavir

SUMMARY:
The purpose of this study is to compare 4 different combinations of anti-HIV drugs and to determine the number of people whose HIV blood levels decrease to 200 copies/ml or less while on the treatment. This study evaluates the safety of these drug combinations, which include an experimental protease inhibitor (PI), amprenavir.

Despite the success that many patients have had with PI treatment regimens, there is still a possibility that patients receiving PIs may continue to have high HIV blood levels. Because of this possibility, alternative drug combinations containing PIs are being studied. It appears that amprenavir, when taken with 3 or 4 other anti-HIV drugs, may be effective in patients with prior PI treatment experience.

DETAILED DESCRIPTION:
A number of studies both within and outside the ACTG have been initiated or are in development to try to address the issue of alternative treatments for patients who either do not achieve or lose virologic control while receiving protease inhibitors (PIs). Amprenavir (APV) is an attractive candidate to investigate as part of salvage regimens because: 1) it has substantial antiretroviral activity; 2) there are preliminary in vitro and in vivo data that suggest that resistance to this agent may be mediated in part by a unique mutation (I50V); and 3) its cross-resistance profile to the approved PIs is uncertain.

Patients are selectively randomized to 1 of 4 study arms based on prior PI experience. Those randomized to Arms A, B, or C receive 2 PIs, 1 of which is amprenavir (APV), and those randomized to Arm D receive a single PI (APV) as part of their treatment regimen, as follows:

Arm A: APV plus saquinavir soft gel capsule (SQVsgc) plus abacavir (ABC) plus efavirenz (EFV) plus adefovir (ADV).

Arm B: APV plus indinavir (IDV) plus ABC plus EFV plus ADV. Arm C: APV plus nelfinavir (NFV) plus ABC plus EFV plus ADV. Arm D: APV plus placebo (NFV, IDV, or SQVsgc) plus ABC plus EFV plus ADV. All patients receive L-carnitine supplementation. All patients receive clinical physical assessments and laboratory testing during study as follows: Weeks 2, 4, and every 4 weeks thereafter. A primary analysis is performed after the last patient has reached 24 weeks. [AS PER AMENDMENT 3/2/00: At that time, all patients are unblinded to their original treatment assignment.] Patients who experience virologic failure are unblinded and may choose 1 of the following 3 options: Continue study medications open-label, permanently discontinue study medications, or selectively continue study medications [AS PER AMENDMENT 3/2/00: from the arm the patient was originally randomized to] and combine with other approved antiretroviral agents. [AS PER AMENDMENT 3/2/00: For patients adding didanosine (ddI) to their regimens, monitoring for the development of pancreatitis is crucial.] Final evaluations are required for those patients who are off drug during the immediate 8-week period following the last dose of study treatment. Beyond 8 weeks, they are followed for incidence of death, cancer, congenital anomalies, and permanent disabilities. [AS PER AMENDMENT 3/2/00: Gilead Sciences has terminated its U.S. development of ADV for HIV infection. Gilead will continue to supply ADV for patients in ACTG 398 until the study closes. Patients who are receiving ADV at the completion of the study may continue to access ADV through the Expanded Access Program, provided that the physician and patient have determined that continued use of ADV is beneficial.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have current virologic failure (2 consecutive HIV blood levels above 1,000 copies/ml) while on PIs.
* Are over 13 years of age (consent of parent or guardian required if under 18).
* Agree to practice abstinence or use effective methods of birth control during the study and for 90 days after.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have hepatitis within 90 days prior to study entry.
* Have a history of a peripheral neuropathy within 60 days of study entry.
* Have an unexplained temperature for a 7-day period.
* Have chronic diarrhea within 30 days prior to study entry.
* Have cancer requiring chemotherapy.
* Received any therapy for infection or other illness within 30 days prior to study entry.
* Have received certain other medications.
* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 475
Dates: Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hammer, Study Chair; John Mellors, Study Chair
Locations (45):
- United States (44):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - USC Univ Hosp & Ambulatory Hlth Care Ctr / USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Emory Hemo Comp Evaluation Clinic / East TN Comp Hemo Ctr, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Tripler Army Med Ctr, Tripler AMC, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med Ctr, Pittsburgh, Pennsylvania
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Pfister M, Labbe L, Hammer SM, Mellors J, Bennett KK, Rosenkranz S, Sheiner LB; Adult AIDS Clinical Trial Group Study 398. Population pharmacokinetics and pharmacodynamics of efavirenz, nelfinavir, and indinavir: Adult AIDS Clinical Trial Group Study 398. Antimicrob Agents Chemother. 2003 Jan;47(1):130-7. doi: 10.1128/AAC.47.1.130-137.2003. PMID 12499180
- [Background] Pfister M, Labbe L, Lu JF, Hammer SM, Mellors J, Bennett KK, Rosenkranz S, Sheiner LB; AIDS Clinical Trial Group Protocol 398 Investigators. Effect of coadministration of nelfinavir, indinavir, and saquinavir on the pharmacokinetics of amprenavir. Clin Pharmacol Ther. 2002 Aug;72(2):133-41. doi: 10.1067/mcp.2002.126183. PMID 12189360
- [Background] Hammer SM, Vaida F, Bennett KK, Holohan MK, Sheiner L, Eron JJ, Wheat LJ, Mitsuyasu RT, Gulick RM, Valentine FT, Aberg JA, Rogers MD, Karol CN, Saah AJ, Lewis RH, Bessen LJ, Brosgart C, DeGruttola V, Mellors JW; AIDS Clinical Trials Group 398 Study Team. Dual vs single protease inhibitor therapy following antiretroviral treatment failure: a randomized trial. JAMA. 2002 Jul 10;288(2):169-80. doi: 10.1001/jama.288.2.169. PMID 12095381
- [Result] Sun J, Nagaraj HN, Reynolds NR. Discrete stochastic models for compliance analysis based on an AIDS Clinical Trial Group (ACTG) study. Biom J. 2007 Aug;49(5):731-41. doi: 10.1002/bimj.200610368. PMID 17726714
- [Result] Ghosh P, Ghosh K, Tiwari RC. Joint modeling of longitudinal data and informative dropout time in the presence of multiple changepoints. Stat Med. 2011 Mar 15;30(6):611-26. doi: 10.1002/sim.4119. Epub 2010 Nov 30. PMID 21337357